CLINICAL TRIAL: NCT00453128
Title: Appraisal of the Diagnostic Rentability of Thorough Analytical Screening Searching Associated Conditions in Patients Newly Diagnosed With Calcium Pyrophosphate Dihydrate Deposition Disease
Brief Title: Diagnostic Rentability of Screening for Associated Conditions in Calcium Pyrophosphate Deposition Disease Patients
Status: Completed | Type: Observational
Sponsor: Sociedade Galega de Reumatoloxía (Other)
Other Study IDs: SGR1
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2007-03-28 (Estimated); Status verified 2007-03

CONDITIONS: Chondrocalcinosis
Keywords: Calcium Pyrophosphate; associated conditions
MeSH Terms: conditions — Chondrocalcinosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether thorough analytical evaluation is useful to diagnose metabolic conditions associated to calcium pyrophosphate deposition disease.

DETAILED DESCRIPTION:
The diagnostic usefulness of screening for hyperparathyroidism, hemochromatosis, hypothyroidism and hypophosphatasia in patients diagnosed with calcium pyrophosphate dihydrate (CPPD) deposition disease is uncertain.

Patients diagnosed with CPPD deposition disease were compared to patients with rheumatoid arthritis and psoriatic arthritis over a 9-year period. All patients were prospectively followed for at least 12 months. Serum calcium, phosphorus, alkaline phosphatase, thyroid-stimulating hormone, ferritin, iron, and total iron binding capacity were determined in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having calcium pyrophosphate dihydrate deposition disease.

Exclusion Criteria:

* Patients mimicking a rheumatoid arthritis disease, with positive rheumatoid factor or with psoriasis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 1997-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José M Pego-Reigosa, MD, PhD, Principal Investigator — Meixoeiro Hospital, Vigo (Pontevedra) SPAIN
Locations (1):
- Meixoeiro Hospital, Vigo, Pontevedra, Spain